CLINICAL TRIAL: NCT04324658
Title: Effect and Tolerance of a Probiotic-based Medical Device (Lactiplus®) Administered to Patients With Irritable Bowel Syndrome
Brief Title: Effect and Tolerance of a Probiotic-based Medical Device Administered to Patients With Irritable Bowel Syndrome
Acronym: Lactiplus
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PIL-DM-L.PLUS-019
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lactiplus — capsules containing L. gasseri LA806

SUMMARY:
This is an observational, open, longitudinal, multicentre study conducted in France.

The study plans to enrol 119 patients with irritable bowel syndrome who will be included by about 50 general practitioners or gastroenterologists consulting in private offices. The treatment, Lactiplus® is a medical device, in the form of capsules containing L. gasseri LA806. The main objective of the study is to assess the effect of a 4-week treatment with the medical device on abdominal pain.

DETAILED DESCRIPTION:
The study is designed as an observational post-market follow-up study, to confirm the performance of the medical device in real life conditions and document its safety profile.

The eligible population corresponds to the population that could benefit from the treatment, according to the MD's instructions for use. Non-inclusion criteria prevent from including patients with other pathologies associated with gastro-intestinal troubles, who may beneficiate from more adequate treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Suffering from IBS (Rome IV criteria), whatever the predominant stool pattern, i.e recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria: Related to defecation; Associated with a change in frequency of stool; Associated with a change in form (appearance) of stool; with symptom onset at least 6 months before diagnosis;
* Having access to electronic tools (computer, tablet…) and an internet connection, allowing him to complete the online self-questionnaire.

Exclusion Criteria:

* Presence of clinical signs of alarm such as rectorrhagia, fever or recent unexpected weight loss or patient with suspicion or evidence of diseases that exclude IBS diagnosis: including but not limited to inflammatory gastrointestinal disease (e.g. Crohn's disease, ulcerative colitis), colorectal cancer, celiac disease, hyperthyroidism, intestinal infection, lactose intolerance, other malabsorption syndromes (e.g.: fructose), bile acid malabsorption;
* History of abdominal surgery except appendectomy;
* Allergy or hypersensitivity to one of the ingredients of the medical device;
* Inability to fill self-questionnaires or to understand the information notice (cognitive or linguistic issues);
* Participation to another clinical study or in the exclusion phase of a previous clinical study;
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with irritable bowel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
assess the effect of a 4-week treatment with the medical device on abdominal pain | 4 weeks

SECONDARY OUTCOMES:
assess the effect of a 4-week treatment with the medical device on digestive troubles | 4 weeks
  global symptom score, intestinal symptoms (discomfort, distension/bloating, urgency to defecate, bowel habit, incomplete rectal emptying), Francis score, Clinical global impression of improvement
assess the effect of a 4-week treatment with the medical device on the patient's quality of life | 4 weeks
assess the effect of a 4-week treatment with the medical device on the patient's intake of treatments (antidiarrheal, antispasmodic, laxative, pro/prebiotics, analgesics) | 4 weeks
assess the tolerance of the medical device | 4 weeks
assess the satisfaction with the medical device | 4 weeks
assess the observance to the treatment and the intake of other medications | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General practitioners or gastroenterologists consulting in french private offices, Paris, France

IPD SHARING:
Plan to Share IPD: No